CLINICAL TRIAL: NCT00674869
Title: Effectiveness of Pit and Fissure Sealants in the Prevention of Dental Caries
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Universitaire de Nice (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 03-APR-12
Record Dates: First submitted 2008-04-22; First posted 2008-05-08 (Estimated); Last update posted 2012-02-22 (Estimated); Status verified 2009-06

CONDITIONS: Caries, Dental
Keywords: sealant; pit; child; over; 6 years old; least
MeSH Terms: conditions — Dental Caries; Van der Woude syndrome | interventions — Pit and Fissure Sealants

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental): pit and fissure sealant on one randomized tooth by pair of permanent molar
  Interventions: Other: pit and fissure sealant
- 2 (No Intervention): No intervention

INTERVENTIONS:
Other: pit and fissure sealant — pit and fissure sealant on one randomized tooth by pair of permanent molar
  Arms: 1

SUMMARY:
This randomized clinical trial is aimed at testing the efficacy of pit and fissure sealants, in a current environmental context different from that of the seventies and eighties. It has a split mouth design. 4OO subjects are included and the duration of follow up is 2 years.

DETAILED DESCRIPTION:
This randomized clinical trial is aimed at testing the efficacy of pit and fissure sealants, in a current environmental context different from that of the seventies and eighties. This study assesses the cost-effectiveness of sealants according to the individual caries risk. This study takes place in Nice, Marseille and Paris (France) and the patients are to be enrolled both in the dental hospitals and in the private practice. In the hospitals, the subjects are recruited directly by the headmasters of the pediatric dentistry or public health departments in the three dental schools. In private practice, the head of the department of pediatric dentistry and / or public health dentistry, of each dental school chooses 4 to 6 private practitioners who are used to place dental sealants in their daily practice. They recruit the subjects among their own patients. The type of study corresponds to randomized clinical trial (Split mouth design) in which the tooth is the statistical unit (one pair of molars considered for each included patient). This study has a direct benefit for individuals. The number of necessary subjects is 328; the sample size is 400. The follow-up duration is 2 years. The treatment is a pit and fissure sealant on one randomized tooth by pair of permanent molars (Split mouth design). Sealant material is set up in accordance with the usual practice of each practitioner. Occlusal exams are conducted every 6 months. The effectiveness of dental sealants and the retention of sealing materials are statistically analyzed according to both the individual caries risk and the clinical protocol

ELIGIBILITY:
Inclusion Criteria:

* child over 6 years old
* patient with at least one carie
* patient with at least one pair of permanent molar: healthy or with equivalent injuries

Exclusion Criteria:

* not cooperating in care
* not speaking french or english

Ages: 6 Years to 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 400 (Actual)
Dates: Start 2004-12; Primary Completion 2008-12 (Actual); Study Completion 2008-12 (Actual)

PRIMARY OUTCOMES:
Caries development | every six month during 2 years

SECONDARY OUTCOMES:
CAOD | every six months during 2 years
Retention sealing of furrows (grooves) | every 6 months during 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Michèle Muller-Bolla, Pr, Principal Investigator — Service d'Odontologie
Locations (1):
- Centre Hospitalier Universitaire de Nice, Nice, France